CLINICAL TRIAL: NCT00908791
Title: An in Vivo Proof of Principle Trial to Determine Whether the Nutritional Supplement Conjugated Linoleic Acid (CLA, Clarinol™) Can Modulate the Lipogenic Pathway in Breast Cancer Tissue
Brief Title: Proof of Principle Trial to Determine if Nutritional Supplement Conjugated Linoleic Acid (CLA) Can Modulate the Lipogenic Pathway in Breast Cancer Tissue
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Lionel.D.Lewis, MD, •Professor of Pharmacology and Toxicology, Geisel School of Medicine, Dartmouth, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D0906
Record Dates: First submitted 2009-05-20; First posted 2009-05-27 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: Conjugated Linoleic Acid; Proof of Principle; Lipogenic Pathway; Clarinol
MeSH Terms: conditions — Breast Neoplasms | interventions — Linoleic Acids, Conjugated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CLA (Experimental): open-label, single-institution proof of principle study of oral CLA in patients with newly diagnosed adenocarcinoma of the breast.
  Interventions: Drug: Conjugated Linoleic Acid (CLA)

INTERVENTIONS:
Drug: Conjugated Linoleic Acid (CLA) — Conjugated linoleic acid (CLA, Clarinol™) oral soft gel capsules will be administered in an open-labeled, manner to all subjects enrolled in the study. Subjects will be treated with 7.5 grams of oral CLA daily, taken in divided dose, twice daily between 8 am and 12 noon and between 8 pm and 12 midnight. CLA will be taken for a minimum of ten days prior to surgical resection of their breast malignancy. In the event that the subject's surgical resection date is delayed, subjects may take CLA for up to 28 days. The last dose of CLA prior to the surgical resection will be taken at 12 midnight or as close as possible to that time and the patient will record the time of the last dosing.
  Other Names: Clarinol

SUMMARY:
Conjugated Linoleic Acid (CLA) is obtained in the human diet by consumption of foods containing ruminant fat. Milk and dairy products have shown the highest amounts of CLA. Clarinol (CLA), is considered a natural supplement and is not regulated by the Food and Drug Administration (FDA). CLA is known to inhibit proliferation of human breast cancer cells and tumors in rodent breast cancer models and reduced Spot 14 (THRSP, S14) and Fatty Acid Synthase (FASN) gene expression in breast cancer cells and tht the two major CLA isomers used in nutritional supplements (C9, t11 and t10, c12) were equipotent in reducing breast cancer cell growth. This study looks at the hypothesis that S14 expression is decreased by CLA and will characterize the major pharmacodynamic (PD) effects of CLA in newly diagnosed Breast cancer patients on Tumor tissue lipogenic pathway. FASN, S14 and Lipoprotein Lipase (LPL), Ki67 and apoptotic index expression will be assessed by quantitative immunohistochemistry (IHC) in initial breast cancer biopsies and compared to that in resected breast tumor tissue after the study subject has been taking CLA for ten to twenty-eight days. Tissue from adjacent breast adipocytes will also be analyzed to determine whether adipose tissue effects can serve as a surrogate marker for those in tumor tissue. A sample of the original biopsy will be compared to the tumor resection sample to determine the levels of CLA in the breast cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* All study patients must have histologically confirmed invasive adenocarcinoma of the breast. Their breast cancer must be resectable clinical stage I or II breast cancer as defined by the current AJCC TNM Staging System (Greene FL, Page DL, Fleming ID, et al.: editors. AJCC cancer staging manual, 6th edition. New York: Springer; 2002).
* All patients must be able to and give informed consent indicating they are aware of the investigational nature of this treatment, prior to entry into the study.
* All subjects must be Age >18 years.
* All subject must have adequate hepatic and renal function documented prior to study entry to include: hepatic transaminases (AST or ALT) ≤ 1.5 times the upper limits of normal, total bilirubin ≤ 1.5 times the upper limits of normal, serum creatinine ≤ 1.5 times the upper limit of normal or eCRCl ≥ 60 mL/min.

Exclusion criteria:

* Patients who have received prior or be receiving radiation therapy for their breast cancer will be excluded.
* Patients who have received prior chemotherapy or receiving chemotherapy or hormonal therapy for their breast cancer will not be included.
* Women must be surgically sterilized or post-menopausal or women of childbearing potential must be using an adequate method of contraception. Women of childbearing potential must be using at least one of the following: oral, implanted, injectable contraceptive hormones, or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or have a partner that is sterile (e.g., vasectomy). Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to start of study therapy. Women who are pregnant or breast-feeding and women of childbearing potential not using an adequate method of birth control will be excluded.
* Patients with gastrointestinal abnormalities including: inability to take oral medication, requirement for intravenous alimentation, or prior surgical procedures affecting nutrient /drug absorption will be excluded.
* A serious uncontrolled medical disorder or active infection which would impair their ability to receive study treatment will be excluded. Significant cardiac disease, including uncontrolled high blood pressure, unstable angina, and congestive heart failure, myocardial infarction within the previous 3 months or serious cardiac arrhythmias will be excluded. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burton L Eisenberg, MD, Principal Investigator — Norris Cotton Cancer Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Norris Cotton Cancer Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women with invasive breast cancer were recruited from the Breast Oncology Clinic at the Norris Cotton Cancer Center at the Geisel School of Medicine at Dartmouth from June 2009 to March 2011. All patients gave written informed consent before entry into the study.
Pre-assignment Details: Participants must have been able to take the study drug for a minimum of 10 days prior to tumor resection. For some potential participants the surgery date was scheduled earlier than 10 days and the study drug was not dispensed.
Groups:
- Conjugated Linoleic Acid: Women with histologically proven invasive non-metastatic breast cancer.
Period: Overall Study
Arm/Group | Conjugated Linoleic Acid
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 24 women completed study treatments. Not all tumors yeiled data for secondary endpoints.
Groups:
- Single Arm Study: Women with histologically proven invasive non-metastatic breast cancer.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.36 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Spot 14 Expression Pre and Post CLA as Assessed by Quantitative Immunohistochemistry and Staining Intensities Scored at 0, 1, or 2
Description: To determine whether ≥ 10 days of CLA consumption suppresses Spot 14 expression in breast cancer tissue in vivo. The staining intensities scoring system used is: no immuostaining (0), weak staining (1), and strong staining (2). The scoring system used objectively and quantitatively assesses the expression of Spot 14, fatty acid synthase, and lipoprotein lipase using the image processing and analysis software Image-Pro Plus™ (MediaCybernetics).
Time Frame: Up to 28 days
Measure: Number; unit: participants
Groups:
- Pre CLA; Post CLA: Women with histologically proven invasive non-metastatic breast cancer.
Arm/Group | Pre CLA | Post CLA
Number analyzed (Participants) | 24 | 24
participants
  Spot 14 Expression Grade 0 | 0 | 0
  Spot 14 Expression Grade 1 | 10 | 22
  Spot 14 Expression Grade 2 | 14 | 2
Statistical Analysis 1: Comparison: Pre CLA vs Post CLA; Test type: Superiority or Other; p = 0.003, McNemar; exact McNemar test for paired binary data

2. Secondary Outcome: Number of Participants With FASN Expression Pre and Post CLA as Assessed by Quantitative Immunohistochemistry and Staining Intensities Scored at 0, 1, or 2
Description: To determine whether ≥ 10 days of CLA consumption suppresses FASN expression in breast cancer tissue in vivo. The staining intensities scoring system used is: no immuostaining (0), weak staining (1), and strong staining (2). The scoring system used objectively and quantitatively assesses the expression of Spot 14, fatty acid synthase, and lipoprotein lipase using the image processing and analysis software Image-Pro Plus™ (MediaCybernetics).
Time Frame: Pre-CLA treatment and up to 2 years Post-CLA treatment
Measure: Number; unit: participants
Arm/Group | Pre CLA | Post CLA
Number analyzed (Participants) | 24 | 24
participants
  FASN Expression Grade 0 | 0 | 0
  FASN Expression Grade 1 | 12 | 14
  FASN Expression Grade 2 | 12 | 10
Statistical Analysis 1: Comparison: Pre CLA vs Post CLA; Test type: Superiority or Other; p = 0.41, McNemar

3. Secondary Outcome: Number of Participants With LPL Expression Pre and Post CLA as Assessed by Quantitative Immunohistochemistry and Staining Intensities Scored at 0, 1, or 2
Description: To determine whether ≥ 10 days of CLA consumption suppresses LPL expression in brest cancer tissue in vivo. The staining intensities scoring system used is: no immuostaining (0), weak staining (1), and strong staining (2). The scoring system used objectively and quantitatively assesses the expression of Spot 14, fatty acid synthase, and lipoprotein lipase using the image processing and analysis software Image-Pro Plus™ (MediaCybernetics).
Time Frame: Pre-CLA treatment and up to 2 years Post-CLA treatment
Measure: Number; unit: participants
Arm/Group | Pre CLA | Post CLA
Number analyzed (Participants) | 24 | 24
participants
  LPL Expression Grade 0 | 4 | 1
  LPL Expression Grade 1 | 16 | 20
  LPL Expression Grade 2 | 4 | 3
Statistical Analysis 1: Comparison: Pre CLA vs Post CLA; Test type: Superiority or Other; p = 0.48, bowker's test of symmetry

4. Secondary Outcome: Number of Participants With Ki67 Expression Pre and Post CLA as Assessed by Quantitative Immunohistochemistry
Description: To determine whether ≥ 10 days of CLA consumption impacts the status of tumor proliferation by calculating the percentage of cells expressing Ki67.
Time Frame: Pre-CLA treatment and up to 2 years Post-CLA treatment
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: Women with histologically proven invasive non-metastatic breast cancer.
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Participants
  Increased expression from Baseline | 5
  Decreased expression from Baseline | 16
Statistical Analysis 1: Comparison: All Study Participants; The Sign-Rank test for paired data; Test type: Superiority or Other; p = 0.029, Sign test

5. Secondary Outcome: Assess Tumor Cell Apoptosis by Immunostaining for Cleaved Caspase 3 Pre and Post CLA
Description: To determine whether ≥ 10 days of CLA consumption impacts the status of tumor cell apoptosis by measuring the presence of immunostaining for cleaved caspase 3.
Time Frame: Pre-CLA treatment and up to 2 years Post-CLA treatment
Measure: Mean (Standard Deviation); unit: stained cells/field
Groups:
- Mean # of Stained Cells Per Microscope Field Pre CLA: Women with histologically proven invasive non-metastatic breast cancer.
Arm/Group | Mean # of Stained Cells Per Microscope Field Pre CLA
Number analyzed (Participants) | 21
stained cells/field
  Mean # of Stained Cells Pre CLA | 1.09 (0.34)
  Mean # of Stained Cells Post CLA | 1.32 (0.34)
Statistical Analysis 1: Comparison: Mean # of Stained Cells Per Microscope Field Pre CLA; Test type: Superiority or Other; p = 0.62, t-test, 2 sided

6. Secondary Outcome: Number of Participants With Measurable Concentration of the Circulating Plasma Free CLA Isomers c9,t11 and t10,c12 Matched to Spot 14 Expression.
Time Frame: Pre-CLA treatment and up to 2 years Post-CLA treatment
Measure: Count of Participants; unit: Participants
Groups:
- Correlation of CLA Isomers Matched to Spot 14 Expression: Number of participants demonstrating a change in concentrations of CLA isomers in correlation to Spot 14 expression.
Arm/Group | Correlation of CLA Isomers Matched to Spot 14 Expression
Number analyzed (Participants) | 21
Participants
  Post-treatment changes | 0
  Incremental changes over baseline | 0
  No correlation | 21
Statistical Analysis 1: Comparison: Correlation of CLA Isomers Matched to Spot 14 Expression; Test type: Superiority or Other; p > 0.05, Other

7. Secondary Outcome: Number of Participants With Measurable Concentration of the Circulating Plasma Free CLA Isomers c9t11 and t10c12 Matched to Ki-67 Expression
Time Frame: Pre-CLA treatment and up to 2 years Post-CLA treatment
Measure: Count of Participants; unit: Participants
Groups:
- Correlation of CLA Isomers Matched to Ki-67 Expression: Number of participants demonstrating a change in concentrations of CLA isomers in correlation to Ki-67 expression.
Arm/Group | Correlation of CLA Isomers Matched to Ki-67 Expression
Number analyzed (Participants) | 21
Participants
  Post-treatment changes | 0
  Incremental changes over baseline | 0
  No correlation | 21
Statistical Analysis 1: Comparison: Correlation of CLA Isomers Matched to Ki-67 Expression; Test type: Superiority or Other; p > 0.05, Other

8. Secondary Outcome: Safety of Short Term Treatment With 7.5 Gram CLA Per Day.
Time Frame: 2 months
Population: Reported toxicities deemed
Measure: Number; unit: participants
Groups:
- # of Grade 1 AEs Deemed "Possibly Related" to CLA; # of Grade 2 AEs Deemed "Possibly Related" to CLA; # of Grade 3 AEs Deemed "Possibly Related" to CLA; # of Grade 4 AEs Deemed "Possibly Related" to CLA: Women with histologically proven invasive non-metastatic breast cancer.
Arm/Group | # of Grade 1 AEs Deemed "Possibly Related" to CLA | # of Grade 2 AEs Deemed "Possibly Related" to CLA | # of Grade 3 AEs Deemed "Possibly Related" to CLA | # of Grade 4 AEs Deemed "Possibly Related" to CLA
Number analyzed (Participants) | 24 | 24 | 24 | 24
participants
  Anorexia | 1 | 0 | 0 | 0
  Constipation | 1 | 0 | 0 | 0
  Diarrhea | 1 | 0 | 0 | 0
  Fatigue | 2 | 0 | 0 | 0
  Headache | 1 | 0 | 0 | 0
  Heartburn | 1 | 0 | 0 | 0
  Insomnia | 1 | 0 | 0 | 0
  Nausea | 2 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: maximum allowed time frames include 4 weeks for screening, 28 days for study drug,and 4 weeks of follow up.
Groups:
- Subjects Taking 1 or More Doses of CLA: Women with histologically proven invasive, non metastatic breast cancer who received at least one day of CLA.
Arm/Group | Subjects Taking 1 or More Doses of CLA
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 14/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Taking 1 or More Doses of CLA (N=24)
abdominal pain (Nervous system disorders) | 1 (5)
alopecia (Skin and subcutaneous tissue disorders) | 1 (3)
Anorexia (Gastrointestinal disorders) | 1 (11)
anxiety (Psychiatric disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (11)
Diarrhea (Gastrointestinal disorders) | 2 (11)
Edema - limbs (Blood and lymphatic system disorders) | 1 (2)
Fatigue (General disorders) | 3 (7)
Headache (Nervous system disorders) | 2 (5)
Heartburn (Gastrointestinal disorders) | 2 (11)
insomnia (General disorders) | 4 (7)
Nausea (Gastrointestinal disorders) | 4 (11)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral Neuropathy (Nervous system disorders) | 2 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (3)
Seroma (Injury, poisoning and procedural complications) | 2 (2)
Elevated WBC (Blood and lymphatic system disorders) | 1 (2)
Skin Infection (Infections and infestations) | 2 (2)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No